CLINICAL TRIAL: NCT03739580
Title: The Comparison of Drug-coated Balloon With Stent Deployment in Popliteal Atherosclerotic Occlusive Lesions
Brief Title: DCB Compared Stenting in Popliteal Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Yong-Quan Gu, Director, vascular suregry department, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DBSP-XWHCMU
Record Dates: First submitted 2018-11-06; First posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Popliteal Stenosis; Popliteal Artery Occlusion; Diabetes
Keywords: drug-coating balloon; stent; popliteal artery; atherosclerotic occlusion
MeSH Terms: conditions — Diabetes Mellitus | interventions — Stents

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- drug-coating balloon (Experimental): drug-coating balloon (Orchid) intervention
  Interventions: Device: DCB angioplasty (Orchid, Acotec Scientific Co. Ltd.)
- stent deployment (Active Comparator): metal bare stent intervention
  Interventions: Device: Stent (Maris,Medtronic.USA or Sinus/Supera, Germany)

INTERVENTIONS:
Device: DCB angioplasty (Orchid, Acotec Scientific Co. Ltd.) — for popliteal stenosis/occlusive lesions, randomised received DCB or Stent deployment.
  Arms: drug-coating balloon
Device: Stent (Maris,Medtronic.USA or Sinus/Supera, Germany) — for popliteal stenosis/occlusive lesions, randomised received DCB or Stent deployment.
  Arms: stent deployment

SUMMARY:
This is a randomized prospective study aiming to compare drug-coated balloons and stent deployment in Popliteal atherosclerotic occlusive lesions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Symptomatic peripheral artery disease:
* Moderate or severe claudication (Rutherford category 2 or 3)
* Critical limb ischemia (Rutherford category 4 or 5)
* Atherosclerotic popliteal artery disease (stenosis > 50%)
* Patients with signed informed consent

Exclusion Criteria:

* Acute critical limb ischemia
* Severe critical limb ischemia (Rutherford category 6)
* Involvement of SFA disease with stenosis
* Continous total occlusion of all proximal infrapopliteal arteries (origin of the anterior tibial artery or tibioperoneal trunk).
* Known hypersensitivity or contraindication to any of the following medications: heparin, aspirin, clopidogrel, or contrast agent
* Age > 80 years
* Severe hepatic dysfunction (> 3 times normal reference values)
* Significant leucopenia, neutropenia, thrombocytopenia, anemia, or known bleeding diathesis
* LVEF < 40% or clinically overt congestive heart failure
* Pregnant women or women with potential childbearing
* Life expectancy <1 year due to comorbidity
* Previous bypass surgery or stenting for the target popliteal artery
* Untreated inflow disease of the ipsilateral pelvic or femoropopliteal arteries (more than 50% stenosis or occlusion)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Primary patency of claudicant patients | 12 months after the index procedure
  Claudicant patients (Rutherford C1-3), primary patency defined as PSVR（peak systolic velocity ratio) ≤2.4, absence of restenosis >50% based on an imaging study (Duplex ultrasound, CT angiography or catheter angiography) at 12 months
Salvage limb rate (for CLI patients) | 12 months after the index procedure
  Limb Salvage is defined as the freedom from secondary major amputation

SECONDARY OUTCOMES:
Rutherford classification | 12 months
ABI | 12 months
  Ankle Brachial index
TcpO2 | 12 months
  transcutaneous oxygen pressure
Wagnar classification | 12 months
  incision healing information of Rutherford C5-6 patients
Target vessel revascularization rate | 12 months
  frequency of repeat intervention or surgical treatment due to loss of patency at the target vessel
Index Limb Ischemia at 12-month Follow up | 12 months
  Index Limb Ischemia is defined by Rutherford/Becker Classification categories 3 through 6.
Major Adverse Events at 12-month Post Procedure | 12 months
  Major adverse events included death, index limb ischemia, index limb amputation, clinically driven target lesion revascularization, and significant embolic events, which were defined as causing end-organ damage.

CONTACTS AND LOCATIONS:
Overall Officials: Yongquan Gu, M.D., Principal Investigator — Xuanwu hospital CMU
Locations (1):
- Gu Yong Quan, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided